CLINICAL TRIAL: NCT00733031
Title: A Phase I, Open-Label, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD6918 Administered Daily as a Single Agent and in Combination Treatment in Adult Patients With Refractory Solid Malignancies
Brief Title: Phase I, Open-label, Dose-escalation, Safety and PK Study of AZD6918
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PK results demonstrate low and variable plasma concentrations so that achieving therapeutic concentrations is unlikely.
Sponsor: AstraZeneca (Industry)
Responsible Party: Judith Ochs, M.D. Medical Science Director, AstraZeneca Pharmaceuticals, LP
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2785C00002
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Cancer,; Solid Tumors; Advanced Solid Malignancies
Keywords: Phase I,; cancer,; solid tumors,; advanced solid malignancies,; dose escalation,; combination treatment,; TRK inhibitor
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- gemcitabine (Experimental): gemcitabine administered in combination with AZD6918
  Interventions: Drug: gemcitabine
- pemetrexed (Experimental): pemetrexed administered in combination with AZD6918
  Interventions: Drug: pemetrexed
- AZD6918 (Experimental): AZD6918 administered alone
  Interventions: Drug: AZD6918

INTERVENTIONS:
Drug: AZD6918 — liquid suspension, daily, oral dose
  Arms: AZD6918
Drug: gemcitabine — intravenous, doses are on an intermittent schedule
  Other Names: Gemzar
  Arms: gemcitabine
Drug: pemetrexed — intravenous, dose administered every 21-days
  Other Names: Alimta
  Arms: pemetrexed

SUMMARY:
The primary purpose of this study is to find out what the maximum tolerated dose is for an experimental drug called AZD6918 based on the side effects experienced by patients with advanced solid malignancies that receive daily AZD6918 alone. It is possible that AZD6918 will be administered twice daily. Then maximum tolerated doses in combination with either gemcitabine or pemetrexed will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors for which standard treatment does not exist or is no longer effective.
* For chemotherapy combination treatment, must be suitable for treatment with either gemcitabine or pemetrexed.
* Relatively good overall health other than cancer.

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells).
* Poor liver or kidney function.
* Serious heart conditions
* History of uncontrolled epilepsy, Parkinson's disease, Alzheimer's disease, brain tumor or any uncontrolled psychiatric or nervous system condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (based on CTCAE version 3.0), laboratory values, vital sign measurements, Karnofsky performance status | Weekly for first two treatment cycles, then every 2-4 weeks

SECONDARY OUTCOMES:
Pharmacokinetic effect of AZD6918 when administered alone and in combination with chemotherapy | According to protocol specified schedule, the number of PK samples collected during Cycle 1 (up to 28 days) based on treatment with AZD6918 alone or in combination with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ochs, MD, Study Director — AstraZeneca; Jeffrey Infante, MD, Principal Investigator — SCRI Development Innovations, LLC; Lia Gore, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Research Site, Aurora, Colorado
  - Research Site, Nashville, Tennessee